CLINICAL TRIAL: NCT01305226
Title: A Prospective Phase III Parallel, Randomised Controlled Trial Using Double-bolus Recombinant Staphylokinase (THR-100) vs Streptokinase in Patients With Acute Myocardial Infarction
Brief Title: A Trial Using Double-Bolus THR-100 Versus Streptokinase
Acronym: THR-100
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bharat Biotech International Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BBIL/STA/05/2007
Record Dates: First submitted 2010-12-28; First posted 2011-02-28 (Estimated); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Acute Myocardial Infarction
Keywords: THR 100
MeSH Terms: interventions — auR protein, Staphylococcus aureus; Streptokinase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Test - THR-100 (Experimental): 120 subjects are to be recruited into the trial, with patients randomized in a 1:1 allocation ratio to THR-100 and Streptokinase 60 subjects are to be recruited into Test arm, and administered 15 mg double-bolus (15mg/15ml), separated by 30 minutes (total 30 mg)
  Interventions: Drug: THR-100
- Streptokinase (Active Comparator): 120 subjects are to be recruited into the trial, with patients randomized in a 1:1 allocation ratio to THR-100 and Streptokinase Streptokinase: Standard regimen (1.5 million IU) is made up in 150 ml of physiological saline or glucose solution and administered intravenously over a period of 60 minutes.
  Interventions: Drug: Streptokinase

INTERVENTIONS:
Drug: THR-100 — THR-100: 15 mg double-bolus (15mg/15ml), separated by 30 minutes (total 30 mg)
  Other Names: Staphylokinase
  Arms: Test - THR-100
Drug: Streptokinase — Streptokinase: Standard regimen (1.5 million IU) is made up in 150 ml of physiological saline or glucose solution and administered intravenously over a period of 60 minutes.
  Other Names: Streptase
  Arms: Streptokinase

SUMMARY:
This novel fibrinolytic agent is a 136 amino acid single chain protein secreted by some strains of Staphylococcus aureus and readily produced by recombinant DNA technology. Two natural variants of recombinant staphylokinase, THR-100 and SakSTAR, have been developed for investigational use in preliminary trials. Like SK, it forms an equimolar complex with plasmin which in turn activates plasminogen to plasmin. Unlike SK, the complexed, activated molecule (which undergoes proteolytic cleavage of the first ten amino acids to generate active staphylokinase) has a high degree of fibrin-selectivity in a human plasma milieu. This fibrin-selectivity is due in large measure to potent activation at the clot surface by trace amounts of plasmin, and rapid inactivation of the circulating complex by antiplasmin. Hence, it provides an interesting and promising alternative therapy.

DETAILED DESCRIPTION:
STUDY SUMMARY/PROTOCOL OUTLINE

Protocol Number: BBIL/STA/O5/2007 Protocol Name: A PROSPECTIVE PHASE III PARALLEL, RANDOMISED CONTROLLED TRIAL USING DOUBLE-BOLUS THR-100 (RECOMBINANT STAPHYLOKINASE) Vs STREPTOKINASE IN PATIENTS WITH ACUTE MYOCARDIAL INFARCTION

Drug under Study: THR-100 (Recombinant Staphylokinase)

Intended Indication: Acute Myocardial Infarction

Study Design: Randomized, Parallel Group, Multicenter and Active-Comparator Trial.

Patient Population: Patients aged 30 to ≤ 75 years presenting with acute myocardial infarction within 12 hours of onset of symptoms presumed secondary to an acute myocardial infarction.

Number of Patients: 120 subjects are to be recruited into the trial, with patients randomized in a 1:1 allocation ratio to THR-100 and Streptokinase over three centers. This sample size of 120 subjects provides power of 0.90 with a significance level of 0.05 to yield a statistically significant early patency difference.

Primary Objectives: To demonstrate efficacy of THR100 as compared with streptokinase by assessment of 12-lead Electrocardiogram, specific cardiac Enzymes levels, pain relief and TIMI-90. (Non-Inferiority study) Secondary Objectives: To evaluate the safety profile of recombinant SAK in comparison with Streptokinase.

Dose Levels: Dose levels (all administered intravenously). THR-100: 15 mg double-bolus (15mg/15ml), separated by 30 minutes (total 30 mg) Streptokinase: Standard regimen (1.5 million IU) is made up in 150 ml of physiological saline or glucose solution and administered intravenously over a period of 60 minutes.

Study Parameters: Primary endpoint:

1. 12-lead Electrocardiogram, ≥50% resolution of ST segment in single ECG lead of maximum deviation present at 90 minutes and 24 hours after start of thrombolytic therapy.
2. Changes in cardiac Enzyme levels of CK-MB and Cardiac Troponin I or T at 6 hrs, 8 hrs, 12-16 hrs and 24 hours after start of thrombolytic therapy.
3. Significant Relief of pain (a 3 point reduction on a 0-5 subjective scale) at end of 2 and 12 hrs after start of thrombolytic therapy. (0-No pain, 1-Slight pain, 2-Mild pain, 3-Moderate pain, 4- Severe pain, 5-Very severe pain).
4. Assessment of culprit coronary vessel patency (TIMI- grade 3) at 90 minutes. (TIMI- Thrombolysis in myocardial infarction). Angiography shall be performed only in patients who fulfil the following guidelines

1. No WPW or LBBB or IV-conduction block or Pacemaker rhythm. 2. ≥0.2 mV ST elevation in ≥2 leads V1-V6 and ≥0.3 mV ST elevation in ≥1 lead V1-V6 3. Sum of ST elevation in V1-V6 plus Sum of ST depression in II, III, aVF ≥0.8 mV (OR)

1. No WPW or LBBB or IV-conduction block or Pacemaker rhythm.
2. ≥0.1 mV ST elevation in ≥2 leads II, III,aVF and ≥0.2 mV ST elevation in ≥1 lead II, III, aVF 5). Sum of ST elevation in I-III, aVF plus Sum of ST depression in V1-V4 ≥0.6 mV.

Secondary endpoints:

Assessment of net clinical benefit, defined as reduced mortality, non-fatal stroke, clinically-evident intracranial hemorrhage, or recurrent myocardial infarction at thirty (30) days.

Assessment of the rates of the following in-hospital events as defined in Appendix 1:

* Heart failure,
* In-hospital death,
* Recurrent myocardial infarction,
* Refractory ischemia,
* need for urgent revascularization,
* Major complications (such as cardiogenic shock, major arrhythmias, pericarditis, tamponade, acute hemodynamically severe mitral regurgitation, acute ventricular septal defect),

Safety considerations:

* Stroke,
* Intracranial hemorrhage (see stroke),
* Major bleeding (other than intracranial hemorrhage),
* Bleeding other than major,
* Serious and non-serious adverse events (see Section 14),
* Allergic reactions,
* Laboratory data. Other angiographic end point CTFC (Corrected TIMI Frame Count), if Angiography performed.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 30 to < 75 years inclusive.
2. Patients presenting within 12 hours with symptoms presumed secondary to an acute myocardial infarction lasting at least 20 minutes and accompanied by ECG evidence of > 1mm of ST elevation in 2 or more limb leads or > 2mm in 2 or more contiguous precordial leads or suspected new left bundle branch block will be eligible.
3. Patients must be in the hospital or the emergency department and able to receive the study medication within 12 hours of onset of symptoms.
4. Females of child-bearing age, not using a generally accepted method of contraception must have a negative urine pregnancy test.
5. Written informed consent should be sought from the patient prior to inclusion in the study. If unable to do so, informed verbal consent will be obtained. If neither is possible, a legally acceptable representative (relative) should provide written consent.
6. NB Verbal or written consent should be followed by written informed consent from the patient at the earliest subsequent opportunity.

Exclusion Criteria:

1. Previous administration of staphylokinase.
2. Active bleeding or known hemorrhagic diathesis.
3. Any history of stroke, transient ischemic attack, dementia, or structural CNS damage e.g. neoplasm, aneurysm, AV malformation.
4. Major surgery or trauma within the past 3 months.
5. Significant hypertension i.e. SBP 180 mm Hg and/or DBP 110 mm Hg at any time from admission to randomization.
6. Current treatment with vitamin K antagonists resulting with an INR > 1.5.
7. Anticipated difficulty with vascular access.
8. Prolonged (>10 min) cardiopulmonary resuscitation or cardiogenic shock.
9. Patients who have participated in an investigational drug study within the past 30 days.
10. Pregnancy or lactation, parturition within the previous 30 days.
11. Any serious concomitant systemic or life limiting disorder that would be incompatible with the trial
12. Patients known to have a history of or life limiting malignant disease or HIV.
13. Significant hepatic or renal dysfunction or any other condition which, in the opinion of the Investigator, makes the patient unsuitable for study entry.
14. Previous participation in this trial

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2010-10; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
To demonstrate efficacy of THR100 as compared with streptokinase by assessment of 12-lead Electrocardiogram, specific cardiac Enzymes levels, pain relief and TIMI-90. (Non-Inferiority study) | up to 4 weeks
  12-lead Electrocardiogram, ≥50% resolution of ST segment in single ECG lead of maximum deviation present at 90 minutes and 24 hours after start of thrombolytic therapy.

SECONDARY OUTCOMES:
To evaluate the safety profile of THR-100 in comparison with Streptokinase | up to 4 weeks
  Assessment of net clinical benefit, defined as reduced mortality, non-fatal stroke, clinically-evident intracranial hemorrhage, or recurrent myocardial infarction at thirty (30) days.

CONTACTS AND LOCATIONS:
Overall Officials: Dr.A Singh, MBBS, MD, Study Director — Bharat Biotech Int. Ltd.
Locations (4):
- India (4):
  - Sri Jayadeva Institute of Cardiology., Bangalore, Karnataka
  - Narayana Hrudayalaya, Bangalore, Karnataka
  - Lotus Super speciality Hospita, Agra, Uttar Pradesh
  - Institute of Post Graduate Medical Education and Research (IPGMER), Kolkata, West Bengal